CLINICAL TRIAL: NCT06650852
Title: A Phase 2 Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Combination Therapy of BRII-179, BRII-835 and Pegylated Interferon Alpha (PEG-IFNα) in Participants With Chronic Hepatitis B Virus (HBV) Infection (ENHANCE)
Brief Title: A Study to Evaluate the Efficacy and Safety of Combination Therapy of BRII-179, BRII-835 and PEG-IFNα in Participants With Chronic Hepatitis B Virus (HBV) Infection (ENHANCE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brii Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRII-179-835-003
Record Dates: First submitted 2024-10-12; First posted 2024-10-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepatitis B Virus (HBV) Infection
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Regimen 1: BRII-179 + BRII-835 + PEG-IFNα (Experimental): Participants will receive BRII-179, BRII-835 and PEG-IFNα as a combination therapy (Regimen 1).
  Interventions: Biological: BRII-179; Drug: BRII-835 (VIR-2218); Biological: PEG-IFNα
- Placebo of BRII-179 + Placebo of BRII-835 + PEG-IFNα (Active Comparator): Participants will receive placebo of BRII-179, placebo of BRII-835 and PEG-IFNα.
  Interventions: Biological: PEG-IFNα; Drug: Placebo of BRII-179; Drug: Placebo of BRII-835
- Regimen 2: BRII-179 + BRII-835 + PEG-IFNα (Experimental): Participants will receive BRII-179, BRII-835 and PEG-IFNα as a combination therapy (Regimen 2).
  Interventions: Biological: BRII-179; Drug: BRII-835 (VIR-2218); Biological: PEG-IFNα

INTERVENTIONS:
Biological: BRII-179 — BRII-179 will be given via intramuscular injection
  Arms: Regimen 1: BRII-179 + BRII-835 + PEG-IFNα; Regimen 2: BRII-179 + BRII-835 + PEG-IFNα
Drug: BRII-835 (VIR-2218) — BRII-835 will be given via subcutaneous injection
  Other Names: elebsiran
  Arms: Regimen 1: BRII-179 + BRII-835 + PEG-IFNα; Regimen 2: BRII-179 + BRII-835 + PEG-IFNα
Biological: PEG-IFNα — PEG-IFNα will be given via subcutaneous injection
  Other Names: Pegylated interferon alfa
Drug: Placebo of BRII-179 — Placebo of BRII-179 will be given via intramuscular injection
  Arms: Placebo of BRII-179 + Placebo of BRII-835 + PEG-IFNα
Drug: Placebo of BRII-835 — Placebo of BRII-835 will be given via subcutaneous injection
  Arms: Placebo of BRII-179 + Placebo of BRII-835 + PEG-IFNα

SUMMARY:
This Phase 2, randomized, double-blind study will evaluate the clinical efficacy and safety of the combination therapy of BRII-179, BRII-835, plus PEG-IFNα compared to PEG-IFNα in adult participants with chronic HBV infection without cirrhosis receiving neucloes(t)ide reverse transcriptase inhibitors (NRTIs) as background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-60 years.
* Body mass index ≥ 18 kg/m2 and ≤ 32 kg/m2.
* Chronic HBV infection for ≥ 6 months.
* On NRTI therapy with HBV DNA < LLOQ for ≥ 6 months.
* Serum ALT and AST ≤ ULN at screening visit.

Exclusion Criteria:

* Any clinically significant chronic medical conditions other than chronic HBV infection that makes the participant unsuitable for participation in the study.
* Significant liver fibrosis or cirrhosis.
* History of clinically significant chronic liver disease from any cause other than chronic HBV infection.
* History of hepatic decompensation.
* Diagnosed or suspected hepatocellular carcinoma.
* Current or past history of infection with HIV, HCV or HDV.
* Any laboratory test abnormality that may contradict treatment with PEG-IFNα.
* Known history of immunological function impairment.
* History of intolerance to intramuscular or subcutaneous injection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants achieving HBsAg seroclearance. | Up to 48 weeks
Percentage of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | Up to 96 weeks

SECONDARY OUTCOMES:
Percentage of participants achieving HBsAg seroconversion. | Up to 48 weeks
Percentage of participants achieving HBsAg seroclearance. | Up to 72 weeks
Percentage of participants achieving HBsAg seroconversion. | Up to 72 weeks
Percentage of participants achieving functional cure. | Up to 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Chen, Study Director — Brii Biosciences Limited
Locations (14):
- China (14):
  - Investigative Site 86001, Beijing, Beijing Municipality
  - Investigative Site 86003, Beijing, Beijing Municipality
  - Investigative Site 86004, Beijing, Beijing Municipality
  - Investigative Site 86005, Beijing, Beijing Municipality
  - Investigative Site 86016, Beijing, Beijing Municipality
  - Investigative Site 86002, Guangzhou, Guangdong
  - Investigative Site 86013, Guangzhou, Guangdong
  - Investigative Site 86015, Shenzhen, Guangdong
  - Investigative Site 86006, Shanghai, Shanghai Municipality
  - Investigative Site 86007, Shanghai, Shanghai Municipality
  - Investigative Site 86010, Chengdu, Sichuan
  - Investigative Site 86011, Chengdu, Sichuan
  - Investigative Site 86012, Chengdu, Sichuan
  - Investigative Site 86009, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No